CLINICAL TRIAL: NCT03104192
Title: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Research Pilot
Brief Title: MOWI Research Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, John A. Batsis, MD, Associate Professor, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: D16182_2; K23AG051681 (NIH)
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Results first posted 2020-07-01 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Obesity
Keywords: frail elderly; telemedicine; obesity; rural health; health promotion; weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Proteins

STUDY DESIGN:
Intervention Model Description: Two Arm Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Develop & Refine MOWI w/o Amulet (2A) (Active Comparator): Develop and refine a mHealth obesity wellness intervention (MOWI) for rural, older, obese adults without the use of Amulet technology.
  Interventions: Behavioral: Develop & Refine MOWI w/o Amulet
- MOWI Weight Loss Maintenance (Experimental): Evaluate the feasibility, acceptability, and potential effectiveness of an 8-session, tri-weekly, psychosocial skills group intervention to support weight loss maintenance post-MOWI.
  Interventions: Behavioral: MOWI Weight Loss Maintenance
- Develop & Refine MOWI w Fitbit (2B) (Active Comparator): Develop and refine a mHealth obesity wellness intervention (MOWI) for rural, older, obese adults with the use of Fitbit technology.
  Interventions: Behavioral: Develop & Refine MOWI w Fitbit
- Develop & Refine MOWI w Fitbit/Protein (2P) (Active Comparator): Develop and refine a mHealth obesity wellness intervention (MOWI) for rural, older, obese adults with the use of Fitbit technology augmented by whey protein.
  Interventions: Dietary Supplement: Develop & Refine MOWI w Fitbit/Protein

INTERVENTIONS:
Behavioral: Develop & Refine MOWI w/o Amulet — The mHealth Obesity Wellness Intervention (MOWI) will be informed by the previous Aim (Aim 1) of this proposal. It will consist of a 12-week, 3x/week program of: weekly nutrition counseling; 2x/week group exercise visits. A dietician and physical therapist will lead the in-person sessions. A wave of 8 individuals each will be assessed at 0, 4, 8 and 12 weeks.
  Other Names: MOWI 2A
  Arms: Develop & Refine MOWI w/o Amulet (2A)
Behavioral: MOWI Weight Loss Maintenance — Participants who successfully completed the initial MOWI program will be offered the opportunity to participate in a 6-month weight management program. This program will consist of 8 group-based skills workshop sessions occurring approximately once monthly (every 3 weeks), which will be 90-120 minutes in length. The overall structure of the program will emphasize the following evidence-based weight management components: Goal setting/action planning, self-monitoring, receiving feedback regarding performance, reviewing relevant goals in the light of feedback, and e. psychological skills for increasing behavioral commitment (acceptance, willingness, thought monitoring, mindful decision making, and values clarification).
  Other Names: MOWI LT
  Arms: MOWI Weight Loss Maintenance
Behavioral: Develop & Refine MOWI w Fitbit — The mHealth Obesity Wellness Intervention (MOWI) will be informed by the previous Aim (Aim 1) of this proposal. It will consist of a 12-week, 3x/week program of: weekly nutrition counseling; 2x/week group exercise visits; and Fitbit to monitor activity. A dietician and physical therapist will lead the in-person sessions. A wave of 8 individuals each will be assessed at 0, 4, 8 and 12 weeks and will also be given Amulet to measure steps, activity type, duration and distance.
  Other Names: MOWI 2B-2
  Arms: Develop & Refine MOWI w Fitbit (2B)
Dietary Supplement: Develop & Refine MOWI w Fitbit/Protein — The mHealth Obesity Wellness Intervention (MOWI) will be informed by the previous Aim (Aim 1) of this proposal. It will consist of a 12-week, 3x/week program of: weekly nutrition counseling; 2x/week group exercise visits; and Fitbit to monitor activity. A dietician and physical therapist will lead the in-person sessions. A wave of 8 individuals each will be assessed at 0, 4, 8 and 12 weeks and will also be given Amulet to measure steps, activity type, duration and distance. We will provide whey protein 3x/week after exercise sessions.
  Other Names: MOWI Protein-2
  Arms: Develop & Refine MOWI w Fitbit/Protein (2P)

SUMMARY:
The goal of this study is to conduct a program of pilot research aimed at developing and evaluating a technology-assisted wellness intervention for older adults with obesity.

DETAILED DESCRIPTION:
The national epidemic of obesity is also affecting older adults, and is associated with an increased risk of disability, nursing home placement and early mortality. Conventional weight loss programs have the potential to reduce body fat, but are difficult to access for older obese adults due to transportation and mobility challenges. The overarching goal of this study is to conduct a program of pilot research aimed at developing and evaluating a technology assisted wellness intervention for older adults with obesity.

Study Timeline:

September 2017 to June 2018:

Goal: Conduct a pilot study of improving weight and physical function in older adults with obesity. An mHealth Obesity Wellness Intervention (MOWI) will integrate Amulet +/- Fitbi with a weekly individual dietician-led nutritional session, along with twice weekly physical therapist led group exercise session.

Participation Duration: Three times weekly for 3 months

ELIGIBILITY:
Inclusion Criteria:

All Aims:

* Age ≥65 years
* Body Mass Index (BMI) ≥ 30kg/m^2
* Waist circumference ≥88cm in females or ≥102cm in males

Aims 2 & 3:

* Have Wi-Fi high speed internet
* Able to obtain medical clearance from doctor
* Have less than a 5% weight loss in past 6 months
* No advanced co-morbidity
* No exercise restrictions
* Not involved in other research studies that may interfere with participation

Exclusion Criteria:

* Severe mental or life-threatening illness
* Dementia
* Substance use
* History of bariatric surgery
* Suicidal ideation
* Unable to perform measures
* Reside in nursing home
* No advanced co-morbidity
* No exercise restrictions
* Not involved in other research studies that may interfere with participation

Aim 4 - had to have completed Aims 2 or 3

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2020-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Batsis, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center / Dartmouth Medical School
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petersen CL, Christensen BC, Batsis JA. Weight management intervention identifies association of decreased DNA methylation age with improved functional age measures in older adults with obesity. Clin Epigenetics. 2021 Mar 2;13(1):46. doi: 10.1186/s13148-021-01031-7. PMID 33653394
- See also: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Qualitative Assessment — https://clinicaltrials.gov/show/NCT03041831
- See also: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Amulet Technology Development & Validation — https://clinicaltrials.gov/show/NCT03085589
- See also: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Home-Based Pilot — https://clinicaltrials.gov/show/NCT03104205

RESULTS

PARTICIPANT FLOW:
Groups:
- MOWI Weight Loss Maintenance: Evaluate the feasibility, acceptability, + potential effectiveness of an 8-session, tri-weekly, psychosocial skills group intervention to support weight loss maintenance post-MOWI.
  MOWI Weight Loss Maintenance: Participants who successfully completed the initial MOWI program will be offered the opportunity to participate in a 6-month weight management program. This program will consist of 8 group-based skills workshop sessions occurring approximately once monthly (every 3 weeks), which will be 90-120 min. The overall structure will emphasize the following evidence-based weight management components: Goal setting/action planning, self-monitoring, receiving feedback regarding performance, reviewing relevant goals in the light of feedback, and e. psychological skills for increasing behavioral commitment.
  Participants in "MOWI Weight Loss Maintenance" were separately enrolled in this Study and did not enter the Maintenance from one or more remaining arms included here.
Period: Overall Study
Arm/Group | Develop & Refine MOWI w/o Amulet (2A) | MOWI Weight Loss Maintenance | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Started | 9 | 27 | 16 | 17
Completed | 9 | 23 | 14 | 14
Not Completed | 0 | 4 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Develop & Refine MOWI w/o Amulet (2A) | MOWI Weight Loss Maintenance | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P) | Total
Number analyzed (Participants) | 9 | 27 | 16 | 16 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (5.1) | 72.7 (4.35) | 73.0 (6.3) | 72.9 (4.4) | 72.5 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 24 | 12 | 14 | 56
  Male | 3 | 3 | 4 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 27 | 16 | 16 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 9 | 27 | 16 | 16 | 68
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 23 | 14 | 14 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Grip Strength
Description: Assessed by a Jamar dynamometer. Sensor-based Thera-bands will measure data on strength change.
Time Frame: Baseline, 12 weeks
Population: For MOWI Weight Loss Maintenance, this was not a measure of evaluation
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Develop & Refine MOWI w/o Amulet (2A) | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 9 | 14 | 14
Kg | 6.2 (5.1) | -2.6 (5.2) | 4.3 (3.4)

2. Primary Outcome: Change in 5 Times Sit-to-Stand (STS)
Description: STS measures lower limb strength (minimal change 2.3 s).
Time Frame: Baseline, 12 weeks
Population: For MOWI Weight Loss Maintenance this was not evaluated
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Develop & Refine MOWI w/o Amulet (2A) | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 9 | 14 | 14
Seconds | -2.9 (2.9) | -1.5 (1.7) | -2.6 (2.2)

3. Primary Outcome: Change in Six-Minute Walk Test (6MWT)
Description: A surrogate for cardiovascular fitness that measures distance (normal 400-700m) related to function. A clinically important difference is 50-55m
Time Frame: Baseline, 12 weeks
Population: For MOWI Weight Loss Maintenance this was not evaluated
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Develop & Refine MOWI w/o Amulet (2A) | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 9 | 14 | 14
Meters | 47.5 (83) | 39.3 (51.6) | 31.8 (27.8)

4. Primary Outcome: Change in Gait Speed (m/s)
Description: Gait speed is measured by the time it takes to walk 20 meters. Gait speed predicts disability and mortality (significant change 0.1 m/s).
Time Frame: Baseline, 12 weeks
Population: For MOWI Weight Loss Maintenance this was not evaluated
Measure: Mean (Standard Deviation); unit: M/s
Arm/Group | Develop & Refine MOWI w/o Amulet (2A) | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 9 | 14 | 14
M/s | 0.2 (0.1) | 0.1 (0.1) | 0.1 (0.1)

5. Primary Outcome: Change in Late-Life Function and Disability Instrument (LLFDI)
Description: LLFDI consists of a 32-item function and 16-item disability (life-task) scales that correlate with gait speed and lower limb function. Higher points indicate better function. Individual raw scores range from 0 to 80, scaled scores are 0 to 100. Each was assessed at baseline and at 12 weeks. We report the differences between baseline/follow-up. Positive score change reflect improved physical function.
Time Frame: Baseline, 12 weeks
Population: For MOWI Weight Loss Maintenance this was not evaluated
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Develop & Refine MOWI w/o Amulet (2A) | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 9 | 14 | 14
Points | 8.6 (8.6) | 9.0 (8.6) | 6.3 (6.9)

6. Secondary Outcome: Change in Behavioral Activation (Patient Activation Measure)
Description: Patient Activation Measure (PAM) assesses knowledge, confidence and skill for managing health and grouped into 4 levels revealing insights into attitudes, motivators, behaviors & outcomes. Higher points indicate better activation. Measures are scored 0-100 units. Scores below reflect changes between baseline and follow-up at 12-weeks. A positive change score indicates improvement in activation
Time Frame: Baseline, 12 weeks post study
Population: For MOWI Weight Loss Maintenance this was not evaluated
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Develop & Refine MOWI w/o Amulet (2A) | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 9 | 14 | 14
Points | 9.2 (11.3) | 18.8 (14.5) | 11.0 (10.8)

7. Secondary Outcome: Change in Subjective Health Status (PROMIS) Physical
Description: Patient Reported Outcomes Measurement Information Systems (PROMIS) Global Short Form. PROMIS is a 10-item instrument capturing physical, mental and social aspects of quality of life having undergone quantitative appraisal and is non-proprietary. Higher points indicate better health. Raw scores are scaled to 0-100. 50 is the mean, 10 points indicates 1 standard deviation. Positive change scores listed below indicate an improvement in subjective health
Time Frame: Baseline, 12-weeks
Population: For MOWI Weight Loss Maintenance this was not evaluated
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Develop & Refine MOWI w/o Amulet (2A) | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 9 | 14 | 14
Points | 3.0 (4.4) | 6.4 (5.3) | 2.3 (3.6)

8. Secondary Outcome: Change in Weight in kg
Description: Change in weight in kg
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Develop & Refine MOWI w/o Amulet (2A) | MOWI Weight Loss Maintenance | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 9 | 14 | 14 | 14
Kg | -4.3 (3.2) | -3.5238 (9.11762) | -5.8 (3.1) | -3.5 (2.9)

9. Secondary Outcome: Change in Waist Circumference in cm
Description: Change in waist and hip circumference in cm
Time Frame: Baseline, 12 weeks post study
Population: For MOWI Weight Loss Maintenance this was not evaluated
Measure: Mean (Standard Deviation); unit: Cm
Arm/Group | Develop & Refine MOWI w/o Amulet (2A) | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 9 | 14 | 14
Cm | -7.6 (4.9) | -6.4 (6.3) | -14.8 (45.5)

10. Secondary Outcome: Average Steps/Expenditure
Description: Average Steps will be measured over a 12 week period
Time Frame: Mean steps over 12 week period of time
Population: For MOWI Weight Loss Maintenance this was not evaluated. For Aim 2A, no fitness device was provided to participants and hence cannot evaluate this outcome in that arm
Measure: Mean (Standard Deviation); unit: Steps
Arm/Group | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14 | 14
Steps | 6494 (3700) | 5127 (3467)

11. Secondary Outcome: Community Healthy Activities Model Program for Seniors Physical Activity Questionnaire (CHAMPS) - Change in Number of Activities
Description: CHAMPS is a self-reported tool in older adults that assesses activity levels and types -
Time Frame: Change Score between baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: activities per week
Arm/Group | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14 | 14
activities per week
  Low intensity activities per week | 3.9 (6.9) | 4.5 (6.9)
  Moderate intensity activities per week | 8.6 (9.2) | 5.2 (9.1)

12. Secondary Outcome: Change in Body Composition - Lean Mass
Description: Lean mass was assessed using bioelectrical impedance for 2P and 2B. This technique was not available for MOWI 2A participants and hence not measured
Time Frame: Baseline, 12 weeks
Population: For MOWI Weight Loss Maintenance this was not evaluated. In 2A (Develop & Refine MOWI w/o Amulet was not measured. This technique was not available for MOWI 2A participants and hence not measured
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14 | 14
Kg | -0.62 (1.4) | -1.44 (1.45)

13. Secondary Outcome: Change in Energy Expenditure
Description: Resting metabolic rate, Change Score (kCal) from Baseline to 12 weeks
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: kCal
Arm/Group | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14 | 14
kCal | -251.6 (579.9) | -206.8 (608.0)

14. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Fasting Plasma Glucose
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14 | 14
mg/mL | -12.2 (25.8) | -4 (13.9)

15. Secondary Outcome: Change in Participant Satisfaction Questionnaire Score
Description: The Participant Satisfaction Questionnaire is a 12-item questionnaire which measures participant satisfaction with intervention participation using a Likert scale (0-5 point scale: very unsatisfied = 0 to very satisfied = 4). Total scores range 0-60: higher scores indicate greater satisfaction with the intervention.Three additional sub-items ask participants to rate their preference for the frequency of sessions, length of group meetings, and total number of group meetings using a Likert scale (-1 - 1 point scale: too few/too short = -1 to 1 = too much/too long). Each of these three items will be interpreted individually and not included in a summed total score. Additionally, this questionnaire includes 1 open-ended response item where participants are asked to leave any additional comments they may have regarding their level of satisfaction with the intervention.
Time Frame: Change score from pre/post (baseline - at end of initial MOWI 12 weeks; follow-up at end of Maintenance study 6 months post-end of MOWI))
Population: only measured in maintenance arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOWI Weight Loss Maintenance
Number analyzed (Participants) | 17
score on a scale | 3.13 (0.773)

16. Secondary Outcome: Change in Credibility and Expectancy Questionnaire Score
Description: The Credibility and Expectancy Questionnaire is a 6-item questionnaire which measures expectancies regarding intervention participation and intervention rationale credibility using a Likert scale (0-10 point scale: responses are anchored to question stems such that, not at all logical/not at all effective/not at all confident/no credibility/not at all comfortable = 0 and very logical/very effective/very confident/high credibility = 10). Total scores range 0-50: higher scores indicate more favorable expectancies regarding participation in the intervention/greater perceived intervention credibility. Additionally, this questionnaire includes 1 open-ended response item that asks participants to leave any additional comments they may have regarding their expectations for the intervention
Time Frame: Baseline (of maintenance intervention) and 6 months (into maintenance) - pre/post
Population: only measured in this intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOWI Weight Loss Maintenance
Number analyzed (Participants) | 17
score on a scale | -0.623529 (2.776583)

17. Secondary Outcome: Community Healthy Activities Model Program for Seniors Physical Activity Questionnaire (CHAMPS) - Change in Number of Not Exercising Activities
Description: CHAMPS is a self-reported tool in older adults that assesses activity levels and types -
Time Frame: Change Score between baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: activities per week
Arm/Group | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14 | 14
activities per week | -3.1 (11.4) | -5.4 (11.6)

18. Secondary Outcome: Community Healthy Activities Model Program for Seniors Physical Activity Questionnaire (CHAMPS) - Change in Duration
Description: CHAMPS is a self-reported tool in older adults that assesses activity levels and types -
Time Frame: Change Score between baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14 | 14
hours
  Not exercising activity duration per week | -2.2 (9.7) | -2.0 (9.0)
  Low intensity activity duration | 1.7 (7.7) | 1.8 (4.9)
  Moderate intensity activity duration | 7.3 (9.6) | 2.4 (7.2)

19. Secondary Outcome: Community Healthy Activities Model Program for Seniors Physical Activity Questionnaire (CHAMPS)
Description: CHAMPS is a self-reported tool in older adults that assesses activity levels and types -
Time Frame: Change in KCal between baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: kCal
Arm/Group | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14 | 14
kCal
  Low intensity caloric expenditure per week | 5.3 (29.5) | 5.7 (19.2)
  Moderate intensity caloric expenditure | 49.4 (74.9) | 13.8 (44.3)

20. Other Pre Specified Outcome: Compliance to Whey Protein Consumption as Measured by Percent of the Total Number of Sessions Whey Could Have Been Taken
Description: Medication adherence, visual analog scale
Time Frame: Baseline, 12 weeks post study
Measure: Number; unit: percentage of total sessions
Arm/Group | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14
percentage of total sessions | 82.6

21. Other Pre Specified Outcome: Change in Food Craving Acceptance and Action Questionnaire Score
Description: The Food Craving Acceptance and Action Questionnaire is a 10-item questionnaire which measures acceptance of food related cravings and urges using a Likert scale (1-7 point scale: never true = 1 to always true = 7). Total scores range 10-70: higher scores indicate greater acceptance of food related cravings and urges.
Time Frame: Change score from pre/post (baseline - at end of initial MOWI 12 weeks; follow-up at end of Maintenance study 6 months post-end of MOWI)
Population: only measured in this arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOWI Weight Loss Maintenance
Number analyzed (Participants) | 17
score on a scale | -1.058824 (6.832556)

22. Other Pre Specified Outcome: Change in Discomfort Intolerance Scale Score
Description: The Discomfort intolerance Scale is a 6-item questionnaire which measures general difficulty managing and regulating physical distress and discomfort using a Likert scale (1-6 point scale: not at all like me = 1 to very much like me = 6). Total scores range 6-36: higher scores indicate greater distress intolerance.
Time Frame: as for outcome 21
Population: only measured in this arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOWI Weight Loss Maintenance
Number analyzed (Participants) | 17
score on a scale | -1.2941 (4.63364)

23. Other Pre Specified Outcome: Change in Physical Activity Acceptance & Action Questionnaire Score
Description: The Physical Activity Acceptance & Action Questionnaire is a 10-item scale which measures acceptance of physical and psychological discomfort in the context of physical activity using a Likert scale (1-7 point scale: never true = 1 to always true = 7). Total scores range 10-70: higher scores indicate greater acceptance of physical and psychological discomfort in the context of physical activity.
Time Frame: as for outcome 21
Population: only measured in this arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOWI Weight Loss Maintenance
Number analyzed (Participants) | 17
score on a scale | 3.2941 (8.54228)

24. Other Pre Specified Outcome: Change in Weight Control Strategies Scale Score
Description: The Weight Control Strategies Scale is a 30-item questionnaire which measures participants' use of behavioral weight control strategies using a Likert scale (1-4 point scale: never = 0 to always = 4). Total scores range 0-120: higher scores indicate greater use of weight control strategies.
Time Frame: as for outcome 21
Population: assessed only in this arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOWI Weight Loss Maintenance
Number analyzed (Participants) | 18
score on a scale | 0.1241 (0.7082)

25. Other Pre Specified Outcome: Change in Voluntary Exercise Questionnaire Score
Description: The Voluntary Exercise Questionnaire is a brief 6-item questionnaire which measures participants' participation in aerobic and strength training activities over the past 3 months and past week. Two items use a Likert scale (1-7 point scale: never = 1 to 7 = very often) and four items ask participants to report frequency of exercise: 0 = 0 days per week to 7 = 7 days per week). Total score range 2-42: Higher scores indicate greater levels of aerobic and strength training activity.
Time Frame: as for outcome 21
Population: only assessed in this arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOWI Weight Loss Maintenance
Number analyzed (Participants) | 18
score on a scale
  Aerobic | -3.1111 (4.523)
  Strength | 0.2222 (3.42234)

26. Other Pre Specified Outcome: Change in Behavioural Regulation in Exercise Questionnaire (BREQ-3) Score
Description: a 24-item assessment of external, introjected, identified, and intrinsic forms of regulation of exercise behavior. Higher scores indicated higher exercise behavior. each is scored on 5 points (0-120). Six subscales - each 4 items (score 0-20 each). A positive change score indicates higher forms of regulation.
Time Frame: as for outcome 21
Population: only assessed in this arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOWI Weight Loss Maintenance
Number analyzed (Participants) | 17
units on a scale
  Amotivation subscale | -0.1324 (0.5312)
  External regulation subscale | -0.3088 (0.7317)
  Introjected regulation subscale | -0.6618 (1.01912)
  Identified regulation subscale | -0.0588 (0.38047)
  Integrated regulation subscale | 0.2794 (0.72824)
  Intrisic motivation subscale | -0.0294 (0.64881)

27. Other Pre Specified Outcome: Change in PROMIS Emotional Distress Short Form Score
Description: an 8 item scale used to measure emotional distress/depression. higher score indicates higher distress. All promis questionnaires raw scores are converted to a scaled score of 0-100. 50 is mean. 10 units on the scale indicate 1 Standard deviation. higher change scores represent reduced emotional distress.
Time Frame: as for outcome 21
Population: Only assessed in this arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOWI Weight Loss Maintenance
Number analyzed (Participants) | 17
units on a scale | 2.8824 (5.20675)

28. Other Pre Specified Outcome: Change in PROMIS Social Isolation Short Form Score
Description: An 8-item scale used to measure perceived social isolation.higher scores indicate higher isolation. All promis questionnaires raw scores are converted to a scaled score of 0-100. 50 is mean. 10 units on the scale indicate 1 Standard deviation. higher change scores represent high isolation.
Time Frame: as for outcome 21
Population: only assessed in this arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOWI Weight Loss Maintenance
Number analyzed (Participants) | 17
units on a scale | -1.5294 (4.30287)

29. Other Pre Specified Outcome: Change in Three Factor Eating Questionnaire Score
Description: 18-item scale measuring eating behavior with 3 subscales (cognitive restraint, emotional eating, uncontrolled eating) using Likert scale (1-4 point scale). Items 1-16 on this scale are reverse scored. The scale score is then entered into the following formula: (cognitive restraint scale score - 3)/9. The outcome is then multiplied by 100. Higher scores indicate higher restraint, emotional eating or uncontrolled eating, respectively. Subscales aretransformed to 0-100 score
  To calculate the emotional eating sub scale, reverse scored items 2, 4, 7, 10, 14 and 16 are summed and then averaged to generate a mean score. The mean score is then multiplied by 6 to generate a scale score. The scale score is then entered into the following formula: (emotional eating scale score - 6)/18. The outcome is then multiplied by 100.
  Positive change scores represent lower restraint, higher emotional eating or higher uncontrolled eating.
Time Frame: as for outcome 21
Population: only assessed in this arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOWI Weight Loss Maintenance
Number analyzed (Participants) | 18
units on a scale
  Uncontrolled eating subscale | -0.823 (14.17778)
  Cognitive restraint subscale | 3.0864 (18.19987)
  Emotional eating subscale | 0.6173 (20.68971)

30. Secondary Outcome: Change in Insulin Level
Description: insulin
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14 | 14
mIU/L | -7.8 (10.1) | -1.32 (4.68)

31. Secondary Outcome: Change in C-peptide
Description: C-peptide
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14 | 14
ng/mL | -0.02 (0.67) | 0.69 (1.25)

32. Secondary Outcome: Change in C-reactive Protein
Description: C-reactive protein
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14 | 14
mg/L | -2.00 (3.96) | -0.65 (1.86)

33. Secondary Outcome: Change in Tumor Necrosis Factor Alpha
Description: tumor necrosis factor alpha
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14 | 14
pg/mL | -0.19 (0.23) | -0.08 (0.28)

34. Secondary Outcome: Change in Interleukin 6
Description: Interleukin 6
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
Number analyzed (Participants) | 14 | 14
pg/mL | 0.10 (2.14) | -0.44 (1.26)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Develop & Refine MOWI w/o Amulet (2A) | MOWI Weight Loss Maintenance | Develop & Refine MOWI w Fitbit (2B) | Develop & Refine MOWI w Fitbit/Protein (2P)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/23 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/23 | 3/14 | 1/14
Other Adverse Events (participants affected / at risk) | 4/9 | 0/23 | 12/14 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Develop & Refine MOWI w/o Amulet (2A) (N=9) | MOWI Weight Loss Maintenance (N=23) | Develop & Refine MOWI w Fitbit (2B) (N=14) | Develop & Refine MOWI w Fitbit/Protein (2P) (N=14)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Temporal Artery biopsy (admission to hospital) for headache
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) — Chest Pain
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Develop & Refine MOWI w/o Amulet (2A) (N=9) | MOWI Weight Loss Maintenance (N=23) | Develop & Refine MOWI w Fitbit (2B) (N=14) | Develop & Refine MOWI w Fitbit/Protein (2P) (N=14)
Cardiovascular (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) — Dyspnea, chest pain
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 10 (17) | 5 (6) — Knee, Hip, neck, shoulder discomofort or any type that impacts joints/muscles
Neurological (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0) | 5 (5) — Headache, TIA, vertigo
Gastrointestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Bloating, diverticulitis
Constitutional (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — fatigue, not feeling well
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Chest cold

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT03104192/Prot_SAP_ICF_000.pdf